CLINICAL TRIAL: NCT06192277
Title: Evaluation of Direct Oral Challenge Clinic in a Rural Ontario Setting - Pilot Project
Brief Title: Evaluation of a Direct Oral Penicillin Challenge in a Rural Community
Acronym: DOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Lisa Allen, Research Coordinator, Director of Reserach, Parry Sound, Huntsville and Bracebridge, Northern Ontario School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: DOC
Record Dates: First submitted 2023-12-15; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Allergy Penicillin
MeSH Terms: interventions — Mass Screening; Penicillins

STUDY DESIGN:
Intervention Model Description: Participants are initially screened to confirm they are at a low risk of reacting to a direct oral penicillin challenge. Low-risk participants are provided oral penicillin and observed for a reaction. If no reaction occurs, (immediate or delayed up to 28 days) patients have their penicillin allergy removed from their electronic medical record with their primary care provider and the local hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low risk (Experimental): Low risk patients will participate in the DOC challenge
  Interventions: Other: Screening; Drug: Low dose Penicillin; Drug: Standard dose Penicillin; Other: Remove allergy label
- High risk (No Intervention): Any participant defined as more than low risk will not receive the DOC

INTERVENTIONS:
Other: Screening — Patients are screened to confirm they are low risk for a penicillin allergy
  Other Names: No treatment
  Arms: Low risk
Drug: Low dose Penicillin — Low risk participants are given a low-dose of oral penicillin followed by 60 minutes of observation
  Arms: Low risk
Drug: Standard dose Penicillin — Participants who have taken the low dose of oral penicillin and have had no reaction are provided a second higher dose of penicillin (250mg) and observed for 60 minutes.
  Arms: Low risk
Other: Remove allergy label — Participants who have no reaction after 28 days have their penicillin allergy label removed from their electronic medical record and hospital record.
  Arms: Low risk

SUMMARY:
This study aims to evaluate the outcomes of a rural-DOC Pilot clinic which will be established in the Huntsville site of Muskoka Algonquin Healthcare. Patients from the Muskoka region who are confirmed to have a low-risk penicillin allergy are eligible for participation in the DOC clinic. Following their experience with the DOC, participation in this study will be voluntary and feedback will be requested from each participant, and local primary care providers. The feedback will be used to assess the impact of the DOC clinic on participants and the medical community over the 2 - year study. Feedback will also be collected to investigate ongoing antimicrobial use for those participants who were successfully delabeled. This will be accomplished by surveying participants at six and twelve months after their DOC.

DETAILED DESCRIPTION:
Penicillin has a well-established role in treating clinical infections in humans and animals. It was the first antibiotic to be mass produced and is still used worldwide. Modifications to the penicillin molecule have yielded derivatives with activity against a broader range of bacteria. However, one of the major limitations to use of penicillin is the incidence of allergic reactions to the drug. Penicillin allergies are reported in more than 10% of outpatients and 15% of inpatients. However, more than 30% of patients have no recollection of the symptoms of their adverse reaction to a medication and the inaccurate or inadequate documentation of adverse reactions can lead to misunderstood allergies. This study will challenge low risk participants to determine if they can safely take penicillin

ELIGIBILITY:
Inclusion Criteria:

* Individuals in the Muskoka region, residing in the catchment area of Muskoka Algonquin Healthcare (Huntsville and South Muskoka site) who meet the following criteria are eligible for the study.

Inclusion Criteria:

* Greater than 18 years of age
* In stable health
* Penicillin allergy that is either self-reported, reported by their primary care provider or previously documented in their electronic medical record
* Successfully screened to ensure they are low-risk for a penicillin allergy and have a PEN-FAST score of <3

Screening Criteria:

* Did not react to penicillin in the past 10 years
* Was never hospitalized with a penicillin reaction
* Have no evidence of a Severe Cutaneous Adverse Reaction (SCAR)
* Have no evidence of a Drug-Related Eosinophilia and Systemic Symptoms (DRESS)
* Have no history of Asthma
* Cannot recall the nature of the penicillin reaction
* Have a history of isolated non-allergic symptoms (eg. GI upset only)
* Only have a family history of penicillin reaction
* If suffer from pruritus (severe itching), with or without maculopapular rash after taking Amoxicillin
* Have no history of IgE mediated hypersensitivity reaction or angioedema

Exclusion Criteria:

* Pregnancy
* Active asthma or any other illness that will increase the participants' risk
* Do not meet the low-risk screening criteria
* Individuals who report an immune-mediated reaction to cephalosporins
* Currently taking Beta Blockers, ACE inhibitors, antihistamines or steroids at a dose greater than prednisone 10mg per day or equivalent
* If study physicians deem them not to be in stable health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Can a DOC operate in a rural community | 1 year
  Report on the number of staff available and who participate, and report on facility availability
Are adequate participants available for DOC | 1 year
  Report on the number of participants who contact the DOC for participation
Can participants be delableled through the DOC | 1 year
  Report on the number of participants who complete the DOC and are delabeled
Number of Reactions | 1 year
  Report on the number and type of reaction. Report the number of participants who are not delabeled.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Wilson, MD, Study Director — Muskoka Algonquin Healthcare
Locations (1):
- Muskoka Algonquin Healthcare, Huntsville, Ontarion, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified study data as requested
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after the study closes for as long as
Access Criteria: Request to PI